CLINICAL TRIAL: NCT05678959
Title: A Three-year, Multi-center, Double-blind, Extension Study to Evaluate the Long-term Safety and Efficacy of Ligelizumab in Patients Who Completed Ligelizumab's Phase III Studies in Food Allergy
Brief Title: Long-term Extension Study of Ligelizumab in Food Allergy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQGE031G12303B; 2022-502366-25-00 (Registry Identifier: EU CTIS)
Record Dates: First submitted 2023-01-09; First posted 2023-01-10 (Actual); Results first posted 2025-10-30 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Food Allergy
Keywords: Food allergy; Peanut allergy; Oral food challenge (OFC); Immunoglobulin E (IgE); ligelizumab
MeSH Terms: conditions — Food Hypersensitivity; Peanut Hypersensitivity | interventions — ligelizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ligelizumab 120 mg (Experimental): Participants received ligelizumab 120 mg and matching placebo (to protect the dose blinding) every 4 weeks.
  Interventions: Drug: Ligelizumab 120 mg
- Ligelizumab 240 mg (Experimental): Participants received ligelizumab 240 mg every 4 weeks.
  Interventions: Drug: Ligelizumab 240 mg

INTERVENTIONS:
Drug: Ligelizumab 120 mg — 1 injection of 1.0 mL ligelizumab and 1 injection of 1.0 mL placebo every 4 weeks
  Arms: Ligelizumab 120 mg
Drug: Ligelizumab 240 mg — 2 injections of 1.0 mL ligelizumab every 4 weeks
  Arms: Ligelizumab 240 mg

SUMMARY:
This was an extension study to evaluate the long-term safety and efficacy of ligelizumab in participants who completed a ligelizumab Phase III study in food allergy.

DETAILED DESCRIPTION:
This was a 3-year extension study with a 16-week follow-up period. The study enabled participants from planned multiple Phase III "core" studies to roll over to this extension study once the participants had completed predefined minimal requirements of a "core" study and agreed to consent to participate in this study.

Participants received ligelizumab treatment allocated in the core study, except for maximum responder (MR) participants performing conditional discontinuation of study treatment. Any participant considered a MR, as defined by an oral food challenge (OFC), performed conditional discontinuation of study treatment. This was to assess whether further treatment was still required because of disease modification by ligelizumab and/or a change in the underlying phenotype following the natural history of the disease (outgrowth of allergy) demonstrated by sustained unresponsiveness.

A subset of participants was offered administration of study treatment at home either by the participant him/herself (self-administration) or by parent/caregiver following training at three visits at the clinic.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed informed consent and or/assent (where applicable) obtained from participant/legal representative prior to enrolling in the rollover study and receiving study medication. If a minor participant providing assent reached the age of legal majority (as defined by local law), he/she was to be re-consented at the next study visit.
* Participants had completed the treatment period in any ligelizumab's Phase III studies in food allergy.
* Participants who were willing to adhere to the study visits and procedures, including receiving injections (study treatment) and participating in the OL-OFC (open label oral food challenge).
* Participants who agreed to continue avoiding exposure to allergens (per core study) and any other foods they were allergic to throughout this study.
* Participants who were able to safely continue into the study as judged by the investigator.

Key Exclusion Criteria:

* Development of a severe or life-threatening episode of an allergic reaction that required intubation and/or intensive care unit (ICU) admission during the core studies.
* Development of a serious adverse event which was suspected to be related to the study treatment judged by the investigator during the core study.
* Development of uncontrolled asthma during the core study that compromised the safety of the participants judged by the investigator.
* Development of clinically significant cardiovascular, neurological, and or psychiatric conditions during the core study that could interfere with or compromise the safety of the participants, interfere with evaluation or interpretation of the study results or preclude completion of the study judged by the investigator.
* Participants who failed to comply with the protocol requirements and procedures during the core study, and in the Investigator's opinion, should not participate in this extension study.
* Platelets <75,000/ul at end of treatment of the core study.

Ages: 6 Years to 57 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 163 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (47):
- United States (25):
  - Allervie Clinical Research, Birmingham, Alabama
  - Allergy and Immunology Associates, Scottsdale, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Allergy and Asthma Associates of Santa Clara Vally Center, San Jose, California
  - Allergy and Asthma Clin Res Inc, Walnut Creek, California
  - UCHealth Outpatient Pavilion, Aurora, Colorado
  - Asthma and Allergy Associates P C, Colorado Springs, Colorado
  - Univ of South Florida Asthma Allergy and Immunology CRU, Tampa, Florida
  - Childrens Healthcare of Atlanta, Atlanta, Georgia
  - Atlanta Allergy and Asthma Clinic, Marietta, Georgia
  - Ann and Robert H Lurie Childs Hosp, Chicago, Illinois
  - Family Allergy and Asthma, Lousiville, Kentucky
  - Johns Hopkins Childrens Center, Baltimore, Maryland
  - Boston Childrens Hospital, Boston, Massachusetts
  - University of Michigan Clinical Trials Office, Ann Arbor, Michigan
  - Respiratory Medicine Research Institute of Michigan, Ypsilanti, Michigan
  - UBMD Pediatrics, Buffalo, New York
  - Northwell Health, New York, New York
  - Mt Sinai Medical Center, New York, New York
  - University Of NC At Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Childrens Hospital MC, Cincinnati, Ohio
  - Childrens Hospital Of Philadelphia, Philadelphia, Pennsylvania
  - Unv of TX Southwestern Medical Center, Dallas, Texas
  - Texas Childrens Hospital, Houston, Texas
  - Seattle Allergy and Asthma Rsch, Seattle, Washington
- Australia (3):
  - Novartis Investigative Site, Brisbane, Queensland
  - Novartis Investigative Site, Parkville, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
- Canada (5):
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
- France (4):
  - Novartis Investigative Site, Angers, France
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Germany (3):
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Berlin
- Novartis Investigative Site, Padua, PD, Italy
- Japan (2):
  - Novartis Investigative Site, Sagamihara, Kanagawa
  - Novartis Investigative Site, Setagaya-ku, Tokyo
- Novartis Investigative Site, Utrecht, Netherlands
- Spain (3):
  - Novartis Investigative Site, Esplugues, Barcelona
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Ghelli C, Costanzo G, Canonica GW, Heffler E, Paoletti G. New evidence in food allergies treatment. Curr Opin Allergy Clin Immunol. 2024 Aug 1;24(4):251-256. doi: 10.1097/ACI.0000000000000999. Epub 2024 May 30. PMID 38814736
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2803
- See also: A Pediatric Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/ppatientsummary/ppatientsummaries?periodicPatientSummaryId=745

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 164 participants were screened in this study, of which one was a screen failure; 163 participants received study treatment.
Period: Overall Study
Arm/Group | Ligelizumab 120 mg | Ligelizumab 240 mg
Started | 81 | 82
Completed | 0 | 0
Not Completed | 81 | 82
Not completed — Study Terminated by Sponsor | 76 | 76
Not completed — Physician Decision | 2 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Guardian Decision | 1 | 0
Not completed — Protocol Deviation | 0 | 1
Not completed — Subject Decision | 1 | 0
Not completed — Technical Problem | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all participants who enrolled into the extension study without screen-failure and who received at least one dose of study treatment during any core study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ligelizumab 120 mg | Ligelizumab 240 mg | Total
Number analyzed (Participants) | 81 | 82 | 163
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.4 (6.95) | 18.9 (6.23) | 19.2 (6.58)
Age, Customized [Number; unit: participants]
  12 - 17 years | 41 | 46 | 87
  18 - 55 years | 40 | 36 | 76
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 36 | 73
  Male | 44 | 46 | 90
Race/Ethnicity, Customized [Number; unit: participants]
  White | 58 | 61 | 119
  Black or African American | 4 | 4 | 8
  Asian | 12 | 10 | 22
  Multiple | 1 | 1 | 2
  Not Reported | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: TEAEs were defined as events where an AE either started after the first dose of extension study treatment and within 16 weeks after the last administered study treatment dose or began prior to the first dose of study treatment but increased in severity (based on preferred term) within 16 weeks after the last study treatment.
Time Frame: Up to approximately 81 weeks
Population: Safety Set 1 included all participants who received at least one dose of study treatment during the extension study.
Measure: Number; unit: percentage of participants
Arm/Group | Ligelizumab 120 mg | Ligelizumab 240 mg
Number analyzed (Participants) | 81 | 82
percentage of participants
  TEAEs | 84.0 | 69.5
  TESAEs | 3.7 | 2.4

2. Secondary Outcome: Number of Participants Tolerating a Single Dose of More Than or Equal to 600 mg of Peanut Protein Without Dose-Limiting Symptoms
Description: Assessed during an open-label oral food challenge (OFC). If missing Week 52-OFC assessments, Week 156-OFC assessments were performed within 380 days (inclusive) after first extension dose date and considered as Week 52-OFC assessments.
Time Frame: Up to approximately 97 weeks
Population: The full analysis set included all participants who enrolled into the extension study without screen-failure and who received at least one dose of study treatment during any core study. Data are reported for participants who responded and had an evaluable value.
Measure: Count of Participants; unit: Participants
Arm/Group | Ligelizumab 120 mg | Ligelizumab 240 mg
Number analyzed (Participants) | 2 | 0
Participants | 1 |

3. Secondary Outcome: Percentage of Participants With TEAEs and TESAEs, Assessed in Participants With at Least One Home Administration of Study Drug
Description: as for outcome 1
Time Frame: Up to approximately 81 weeks
Population: Safety Set 1 included all participants who received at least one dose of study treatment during the extension study. Number analyzed is the number of participants with available data.
Measure: Number; unit: percentage of participants
Arm/Group | Ligelizumab 120 mg | Ligelizumab 240 mg
Number analyzed (Participants) | 36 | 46
percentage of participants
  TEAEs | 86.1 | 67.4
  TESAEs | 5.6 | 0

4. Secondary Outcome: Change From Baseline in Total Scores in the Food Allergy Quality of Life Questionnaire (FAQLQ) Teenager Form (FAQLQ-TF)
Description: The FAQLQ-TF is a self-reported instrument designed for adolescents aged 13-17 to assess the impact of food allergy on health-related quality of life (HRQoL). The questionnaire includes three domains (emotional impact, allergen avoidance and dietary restrictions, and risk of accidental exposure). Each item was scored on a 7-point scale, with a higher score indicating greater impairment in HRQoL. The total score was calculated as the arithmetic average of all completed items. The possible range for the total score was 1 (minimum) to 7 (maximum). The higher the score, the greater the impairment in HRQoL. OFC = oral food challenge.
Time Frame: Up to approximately 97 weeks
Population: The full analysis set included all participants who enrolled into the extension study without screen-failure and who received at least one dose of study treatment during any core study. Only participants with a value at both the baseline and post-baseline visits were included.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Ligelizumab 120 mg | Ligelizumab 240 mg
Number analyzed (Participants) | 0 | 1
Unit on a scale |  | 1.13 (NA) — Standard deviation was not calculable due to the single data point.

5. Secondary Outcome: Change From Baseline in Total Scores in the Food Allergy Quality of Life Questionnaire (FAQLQ) Adult Form (FAQLQ-AF)
Description: The FAQLQ-AF is a self-reported instrument designed for adults aged 18-55 to assess the impact of food allergy on health-related quality of life (HRQoL). The questionnaire includes four domains (emotional impact, allergen avoidance and dietary restrictions, risk of accidental exposure, and food allergy-related health). Each item was scored on a 7-point scale, with a higher score indicating greater impairment in HRQoL. The total score was calculated as the arithmetic average of all completed items. The possible range for the total score was 1 (minimum) to 7 (maximum). The higher the score, the greater the impairment in HRQoL. OFC = oral food challenge.
Time Frame: Up to approximately 97 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Ligelizumab 120 mg | Ligelizumab 240 mg
Number analyzed (Participants) | 4 | 2
Unit on a scale | 0.32 (0.873) | 0.29 (1.048)

6. Secondary Outcome: Change From Baseline in Total Scores in the Food Allergy Independent Measure (FAIM) Teenager Form (FAIM-TF)
Description: The FAIM-TF is a self-reported instrument designed for adolescents aged 13-17. It aims to reflect the participant's perceived food allergy severity and food allergy-related risk. The questionnaire consists of six questions. The first four questions assess the participant's food allergy expectation outcomes, and the remaining two questions reflect aspects of the perceived severity of food allergy. The total score was calculated as the arithmetic average of all completed items. The possible range for the total score was 1 (minimum) to 7 (maximum). The higher the score, the greater the perceived risk or chance of adverse events occurring. OFC = oral food challenge.
Time Frame: Up to approximately 97 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Ligelizumab 120 mg | Ligelizumab 240 mg
Number analyzed (Participants) | 0 | 1
Unit on a scale |  | 0.33 (NA) — Standard deviation was not calculable due to the single data point.

7. Secondary Outcome: Change From Baseline in Total Scores in the Food Allergy Independent Measure (FAIM) Adult Form (FAIM-AF)
Description: The FAIM-AF is a self-reported instrument designed for adults aged 18-55. It aims to reflect the participant's perceived food allergy severity and food allergy-related risk. The questionnaire consists of six questions; The first four questions assess the participant's food allergy expectation outcomes, and the remaining two questions reflect aspects of the perceived severity of food allergy. The total score was calculated as the arithmetic average of all completed items. the range for each item and the total score is from 1 (minimum) to 7 (maximum). The possible range for the total score was 1 (minimum) to 7 (maximum). The higher the score, the greater the perceived risk or chance of adverse events occurring. OFC = oral food challenge.
Time Frame: Up to approximately 97 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Ligelizumab 120 mg | Ligelizumab 240 mg
Number analyzed (Participants) | 3 | 2
Unit on a scale | -0.44 (0.385) | 0.42 (1.296)

8. Secondary Outcome: Change From Baseline in the Medical Outcomes Study 36-item Short Form Version 2 Acute Version (SF-36v2) Physical Component Score (PCS) and Mental Component Score (MCS)
Description: The SF-36v2 Health Survey is a 36-item instrument that measures generic health-related quality of life. It contains 8 scales and 2 component summary indices evaluating physical, social, and emotional functioning in addition to general health perceptions and mental health. PCS and MCS scores range from 0 to 100, with higher scores indicating better health outcomes.
Time Frame: Up to approximately 97 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Ligelizumab 120 mg | Ligelizumab 240 mg
Number analyzed (Participants) | 3 | 2
Unit on a scale
  PCS | 0.3 (5.03) | 7.0 (11.31)
  MCS | 0.0 (6.00) | -13.0 (21.21)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 16 weeks post treatment, up to a maximum duration of approximately 81 weeks.
Arm/Group | Ligelizumab 120 mg | Ligelizumab 240 mg
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/82
Serious Adverse Events (participants affected / at risk) | 3/81 | 2/82
Other Adverse Events (participants affected / at risk) | 47/81 | 43/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ligelizumab 120 mg (N=81) | Ligelizumab 240 mg (N=82)
Cardiomyopathy (Cardiac disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Swollen tongue (Gastrointestinal disorders) | 1 | 0
Swelling face (General disorders and administration site conditions) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus allergic (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ligelizumab 120 mg (N=81) | Ligelizumab 240 mg (N=82)
Injection site erythema (General disorders and administration site conditions) | 7 | 14
Injection site induration (General disorders and administration site conditions) | 1 | 6
Injection site oedema (General disorders and administration site conditions) | 4 | 11
Injection site swelling (General disorders and administration site conditions) | 2 | 7
COVID-19 (Infections and infestations) | 6 | 7
Gastroenteritis (Infections and infestations) | 2 | 6
Influenza (Infections and infestations) | 9 | 4
Nasopharyngitis (Infections and infestations) | 19 | 17
Upper respiratory tract infection (Infections and infestations) | 12 | 10
Viral infection (Infections and infestations) | 5 | 3
Headache (Nervous system disorders) | 13 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2023-08-14): https://cdn.clinicaltrials.gov/large-docs/59/NCT05678959/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-15): https://cdn.clinicaltrials.gov/large-docs/59/NCT05678959/SAP_001.pdf